CLINICAL TRIAL: NCT06665919
Title: Randomized Controlled Trial for Evaluating CYP2C19 Allele Genotype-guided Clopidogrel Treatment Outcomes in Real-world Practice After the ePCI
Brief Title: The Study of CYP2C19 Genotype-Guided Clopidogrel Treatment Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vistamedi Ltd. (Industry)
Collaborators: Tbilisi State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BREC-TSMU#2-2023/103
Record Dates: First submitted 2024-09-29; First posted 2024-10-30 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Clopidogrel Resistance; Coronary Thrombosis; Adverse Cardiac Events; Bleeding; Hospitalisations; Death; Death From Cardiovascular Disease
Keywords: CYP2C19 Genotype-guided antiplatelet treatment; Clopidogrel Resistance; Double Antiplatelet Treatment; Chronic Coronary Artery Disease; Implementation of Genotype-guided Medication Treatment; Outcome Study
MeSH Terms: conditions — Coronary Artery Disease; Coronary Thrombosis; Cardiovascular Diseases; Hemorrhage; Death

STUDY DESIGN:
Intervention Model Description: To evaluate CYP2C19 allele genotype-guided clopidogrel treatment outcomes after the ePCI study participants were randomly allocated into parallel study arms. Experimental arm participants have undergone CYP2C19 genotyping. Carriers of normal *2, *3 alleles - "normal metabolizers" phenotype separated as the experimental arm and participants randomly allocated in the comparators arm without CYP2C19 genotyping - the "unspecified metabolizers" phenotype, have been intervened with clopidogrel-based preventive antiplatelet treatment. Carriers of LoF *2, *3 alleles - the "poor metabolizers" phenotype, have been separated in the experimental arm, assigned as the additional comparators and intervened with preventive antiplatelet treatment alternative to clopidogrel. Clinical and non-clinical outcome measures are expected to be compared between parallel study groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal Metabolizers of Clopidogrel (Experimental): 157 study participants diagnosed with chronic coronary artery disease who had undergone elective PCI, tested with CYP2C19 genotyping and identified as NFA *2, *3 carriers.
  Interventions: Other: CYP2C19 Genotype-Guided Clopidogrel Treatment
- Passive Metabolizers of Clopidogrel (Experimental): 43 study participants diagnosed with chronic coronary artery disease who had undergone elective PCI, tested with CYP2C19 genotyping, identified as LoF *2, *3 alleles carriers.
  Interventions: Other: CYP2C19 Genotype Guided Antiplatelet Treatment Alternative to Clopidogrel
- Unspecified Metabolizers of Clopidogrel (Active Comparator): 83 participants diagnosed with chronic coronary artery disease who had undergone elective PCI were allocated to the arm through the randomization, without CYP2C19 genotyping and clopidogrel metabolism phenotype have not been specified.
  Interventions: Other: The Conventional Clopidogrel Treatment

INTERVENTIONS:
Other: CYP2C19 Genotype-Guided Clopidogrel Treatment — Clopidogrel as a component of preventive antiplatelet treatment such as double antiplatelet treatment (DAPT), or an antiplatelet drug (clopidogrel) combined with the non-vitamin K antagonist oral anticoagulants (NOAC), incl. triple antiplatelet treatment (Aspirin, Clopidogrel and a NOAC), or antiplatelet monotherapy (Clopidogrel).
  Arms: Normal Metabolizers of Clopidogrel
Other: CYP2C19 Genotype Guided Antiplatelet Treatment Alternative to Clopidogrel — An antiplatelet drug alternative to clopidogrel in conventional dosing regimen, as a component of preventive antiplatelet treatment, such as double antiplatelet treatment (DAPT) with ticagrelor or prasugrel, or prasugrel combined with the non-vitamin K antagonist oral anticoagulants (NOAC), or antiplatelet monotherapy (ticagrelor, or prasugrel).
  Arms: Passive Metabolizers of Clopidogrel
Other: The Conventional Clopidogrel Treatment — Clopidogrel as a component of preventive antiplatelet treatment such as double antiplatelet treatment (DAPT), or clopidogrel combined with the non-vitamin K antagonist oral anticoagulants (NOAC), incl. triple antiplatelet treatment (Aspirin, Clopidogrel and a NOAC), or antiplatelet monotherapy (Clopidogrel).
  Arms: Unspecified Metabolizers of Clopidogrel

SUMMARY:
The study purposed to learn how clopidogrel-based antiplatelet treatment for preventing adverse cardiovascular events after ePCI works in chronic coronary artery disease when guided by personal genetic characteristics for drug metabolism.

The study aimed to answer two research questions:

* Does CYP2C19 genotype-guided clopidogrel treatment provide better clinical outcomes when compared with conventional treatment selection led without CYP2C19 genotyping?
* Can CYP2C19 genotype-guided antiplatelet treatment be beneficially applied in real-world clinical practice?

After obtaining the informed consent eligible study participants screened by inclusion and exclusion criteria were randomized and allocated into two groups:

* for whom the CYP2C19 genotype-guided clopidogrel treatment has been applied - the experimental group,
* for whom conventional clopidogrel has been applied without CYP2C19 genotyping - the control group.

The experimental group participants underwent CYP2C19 genotyping. Study participants with CYP2C19 normal function alleles (NFA) *2, *3 genotypes constituted the separate experimental arm and received clopidogrel-based preventive antiplatelet treatment.

Participants with CYP2C19 *2 and *3 loss of function (LoF) alleles were allocated to the separate experimental group and received preventive antiplatelet treatment alternative to clopidogrel.

Study participants who had not undergone CYP2C19 genotyping and received conventional preventive antiplatelet treatment with clopidogrel were assigned as active comparators.

All participants in the experimental and comparator groups underwent standard clinical investigations by current guideline recommendations for:

* the initial assessment,
* follow-up and detection of major adverse cardiovascular events. All patients received the conventional drug treatment by current guideline recommendations for chronic coronary artery disease and comorbid condition management and adverse cardiovascular events prevention.

The main research outcome measures include:

* evaluating clinical outcomes of CYP2C19 genotype-guided antiplatelet treatment application,
* describing models for application of CYP2C19 genotype-guided antiplatelet treatment,
* learning about potential access points to the real practice process pipeline for implementation of genotype-guided medication treatment.

DETAILED DESCRIPTION:
The concept of the study is based on current evidence from multiple genetic and clinical studies. At this stage of development preventive treatment of chronic coronary artery disease after ePCI is challenged by risks related to multi-morbidity, recurrent MACCEs and bleeding. Scientific evidence broadly supports pharmacogenetic approaches for routine use of P2Y12 inhibitors (clopidogrel or alternative). Clopidogrel remains the most commonly used P2Y12 inhibitor in the post-ePCI settings. Along with disease-related and co-morbid factors treatment effects are influenced by the variability of the CYP2C19 genotype in the population, which significantly increases the risk of MACCE in loss of function allele (LoF) carriers even with conventional clopidogrel treatment. To improve treatment, a pharmacogenetic expediency model for drug selection is introduced. CYP2C19 allele genotype-guided clopidogrel or an alternative P2Y12 inhibitor treatment is based on robust evidence.

The study aimed to learn the comparative benefits of CYP2C19 genotype-guided versus conventional clopidogrel treatment selection applied in real clinical practice for preventing adverse cardiovascular events after ePCI in chronic coronary artery disease.

For this purpose, the randomized parallel-group controlled study for CYP2C19 genotype-guided clopidogrel treatment outcomes evaluation for chronic coronary artery disease after the ePCI in real-world practice was conducted.

The study addressed research-specific objectives:

* forming and random allocating of participants into study arms for CYP2C19 allele genotype-guided versus conventional clopidogrel treatment,
* ensuring RT-PCR based assay for CYP2C19 *2, *3 LoF alleles detection in randomly selected study participants and forming the experimental study groups,
* characterizing clinical traits of study participants and observing adverse clinical events during the 12-month course of study intervention treatment;
* evaluating the clinical and non-clinical study outcomes. Following the completion of the informed consent, 283 patients eligible for inclusion and exclusion criteria have been enrolled in the study and randomly allocated into two groups.

  83 participants created the control group. They did not undergo CYP2C19 genotyping and received conventional antiplatelet treatment based on clopidogrel.

  200 participants were tested for CYP2C19 *2, *3 allele genotype. 157 of those who revealed normal CYP2C19 *2, *3 allele genotype received conventional preventive antiplatelet treatment based on clopidogrel and created a separate experimental arm.

  43 participants who revealed CYP2C19 *2, *3 LoF allele genotype required preventive antiplatelet treatment alternative to clopidogrel - based on ticagrelor or prasugrel were allocated into another separate experimental arm and assigned as the perspective arm for further study.

Before inclusion, informed consent was obtained from all study participants (or their legal representatives).

The randomization and study arm allocation processes were blinded for participants, healthcare teams providing medical care and study outcomes assessors. Nevertheless, after randomization and genetic testing, CYP2C19 allele genotyping results were disclosed to the medical care team and study participants to make ongoing clinical management safe and transparent but remained blinded for study outcomes assessors.

RT-PCR-based laboratory assay for CYP2C19 *2, *3 alleles genotyping was carried out only once after randomization for each study participant allocated into the experimental group. Tests were performed in the diagnostic laboratory of Vistamedi Ltd served as the central study laboratory.

The laboratory test report was provided to the authenticated investigator and as well as participant and entered in the study data report form.

Regular healthcare teams conducted clinical management of study participants in a real practice environment including medication treatment under conventional guideline recommendations were detected and initially reported major adverse cardiovascular outcomes, other adverse events, or additional clinical conditions diagnosed or study-related circumstances emerged through the study follow-up period up to the end of the study. Study participants (or their legal representatives) were also allowed to report adverse clinical outcomes, events or emerging circumstances.

For a study participant, the expected end of the study is defined as the end date of the 12-month follow-up from the date of the index ePCI. However, in the case of the clinical endpoint which corresponded to and defined the study outcome measure, the date of such endpoint event was determined as the end of the study, even if earlier than 12 months from the index ePCI.

The study participant could terminate participation by his or her independent decision, from any time of the research and for any reason, which could or could not be established.

Early withdrawal of a participant from the study was considered reasonable if there was repeated non-adherence to the treatment of study interest, rather than sporadic, or when there was preferred to terminate treatment based on the justified best interests of the participant.

Clinical outcomes conventionally defined by the Standardized Data Collection for Cardiovascular Trials Initiative (SCTI), the US Food and Drug Administration (FDA), the Academic Research Consortium for High Bleeding Risk (ARC-HBR) and WHO have been measured by clinical endpoints developed over the course of clinical cases.

Certain elements of the Coronary Revascularization Outcome Questionnaire (CROQ) and Patient-Reported Outcomes Measurement Information System®-Plus-Heart Failure profile were used for measuring of Patient-Reported Outcomes (PROs).

Study results were also analyzed using other non-clinical outcome measures that characterized the effectiveness of СYP2C19 genotype-guided P2Y12 inhibitor treatment utilization in real practice.

Data from each study participant were entered into a CRF, the form of which was the same for all participants and study centers.

Study data are collected, stored, and processed into a custom-designed electronic database. Identifiers, study variables and record data are validated with codes to ensure personal data protection.

Personal data, code keys and definitions, and research data are warehoused in separate databases. Only authenticated researchers have access to them. Research data collection centers do not have an internet connection or any other access to the database files.

Study data processing is only allowed by the study procedures given in the study protocol.

After the data collection, the database containing the personal data of the study participants will be deleted.

The de-identified electronic database will be stored after the end of the study for further research purposes for an indefinite period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic coronary artery disease;
* Undergone elective PCI within the last 12 weeks without procedure-related complications;
* LVEF≥38% after index PCI;
* Completed informed consent form for participation in the study;

Exclusion Criteria:

* Concomitant using of potent CYP3A4 or CYP2C19 inhibitors;
* Morbid obesity, BMI 40 kg/sq.m or more;
* Type 1 diabetes mellitus;
* Poorly controlled type 2 diabetes mellitus, HbA1c - 9% or more;
* Acute Myocardium Infarction;
* Coronary artery bypass grafting performed within the last 12 weeks;
* Valvular heart disease due to dysplasia, connective tissue disorders or inflammatory disorders, or valvular disorders requiring cardiac surgery;
* History of severe hepatic impairment;
* Severe chronic kidney disease;
* Clinically important leucopenia, lymphopenia, thrombocytopenia or thrombocytosis;
* History of hemorrhagic diathesis or coagulopathy;
* An active or an obvious threat of bleeding (including GI bleeding):
* Bleeding within the past 6 months that required hospitalization;
* Blood transfusion during the past 6 months or its refusal;
* History of intracranial hemorrhage;
* Cardiac or non-cardiac degenerative disease, including: cardiomyopathy, restrictive lung disease, or Neurodegenerative diseases;
* Malignant tumor (cancer) that limits life expectancy to less than one year;
* Current chemotherapy or immunosuppressive therapy;
* Ongoing immunosuppression or immunosuppressive conditions;
* Pregnancy or lactation period;
* Any disease/condition control of which is not achieved;
* Personal (patient/physician dependent) or health care system-related circumstances that can restrict or limit any study procedures or operations.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Levan Jijeishvili, MD, MPH, Study Director — Vistamedi Ltd., Tbilisi Georgia; Konstantine Liluashvili, MD., PH.D., Principal Investigator — Tbilisi State Medical University; Tornike Batavani, MD, MPH, Study Chair — Vistamedi Ltd. Tbilisi, Georgia
Locations (4):
- Georgia (4):
  - 1st University Clinic of the Tbilisi State Medical University, Tbilisi
  - Cardio Expert Ltd., Clinic Cardio, Tbilisi
  - T. Oragvelidze Cardiology Center, Tbilisi
  - Tbilisi Institute of Medicine, Tbilisi

IPD SHARING:
Plan to Share IPD: Yes
After deidentification of the data records, the deidentified IPD used for the results section intended for article publication will be shared.
  The data set will contain certain demographics, risk factors, cardiovascular morbidity, co-morbidity, coronary angiography, doppler-echocardiography, medication selection records of intervention and control group patients as well as CYP2C19 gene *2, *3 allele profile of the intervention group patients.
  Meta-data in the form of tables, figures, text or appendices will be available as well.
  The study protocol, variable and recorded data coding, statistical analysis plan and informed consent form will be shared as well.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will be available 1 month following the publication of the article containing study results. The anticipated date of final data collection for the primary outcome measures is March 2025. At this time two manuscripts for publication submission are expected to be completed and the study IPD will be available for sharing.
  Before this time supporting information will be shared. After sharing IPD, supporting information will be available for researchers in the field related to this study.
  The study IPD will remain available for sharing 36 months after the article publication.
Access Criteria: IPD and supportive information will be accessible for researchers and investigators who will provide a methodologically sound proposal and whose proposed use of the data will be approved by the independent review and ethics boards. The proposal should display aims and types of IPD analysis, show intentions for IPD meta-analysis.
  Possibility and appropriateness of the IPD for sharing should be confirmed by the National Personal Data Protection Service of Georgia.
  The proposal can be submitted up to 36 months following the study article publication. After 36 months the IPD will be available in the VistaMedi Ltd data warehouse but without investigators support other than deposited meta-data.
  Information regarding proposal submitting, IPD accessing procedures and more detailed plan for sharing IPD, Study Protocol, Statistical Analysis Plan (SAP), Informed Consent Form (ICF) and Variable Data codes will be released on the VistaMedi Ltd official website http://vistamedi.ge/en/.

REFERENCES:
- [Background] Timmis A, Vardas P, Townsend N, Torbica A, Katus H, De Smedt D, Gale CP, Maggioni AP, Petersen SE, Huculeci R, Kazakiewicz D, de Benito Rubio V, Ignatiuk B, Raisi-Estabragh Z, Pawlak A, Karagiannidis E, Treskes R, Gaita D, Beltrame JF, McConnachie A, Bardinet I, Graham I, Flather M, Elliott P, Mossialos EA, Weidinger F, Achenbach S; Atlas Writing Group, European Society of Cardiology. European Society of Cardiology: cardiovascular disease statistics 2021. Eur Heart J. 2022 Feb 22;43(8):716-799. doi: 10.1093/eurheartj/ehab892. PMID 35016208
- [Background] N. Mikaia, L. Jijeishvili, K. Liluashvili, M. Sebiskveradze, Z. Kavtaria, L. Bakashvili, M. Okujava, Implementation of molecular markers targeting thrombosis-related conditions in the real clinical practice, Clinica Chimica Acta, Volume 558, Supplement 1, 2024, 119263, ISSN 0009-8981, https://doi.org/10.1016/j.cca.2024.119263. (https://www.sciencedirect.com/science/article/pii/S0009898124015043)
- [Background] Zhang Y, Shi XJ, Peng WX, Han JL, Lin BD, Zhang R, Zhang YN, Yan JL, Wei JJ, Wang YF, Chen SW, Nan N, Fang ZW, Zeng Y, Lin Y. Impact of Implementing CYP2C19 Genotype-Guided Antiplatelet Therapy on P2Y12 Inhibitor Selection and Clinical Outcomes in Acute Coronary Syndrome Patients After Percutaneous Coronary Intervention: A Real-World Study in China. Front Pharmacol. 2021 Jan 20;11:582929. doi: 10.3389/fphar.2020.582929. eCollection 2020. PMID 33551797
- [Background] Beitelshees AL, Stevenson JM, El Rouby N, Dillon C, Empey PE, Fielstein EM, Johnson JA, Limdi NA, Ong HH, Franchi F, Angiolillo DJ, Peterson JF, Rosenman MB, Skaar TC, Tuteja S, Cavallari LH; IGNITE Pharmacogenetics Working Group. Evaluating the extent of reusability of CYP2C19 genotype data among patients genotyped for antiplatelet therapy selection. Genet Med. 2020 Nov;22(11):1898-1902. doi: 10.1038/s41436-020-0894-2. Epub 2020 Jul 17. PMID 32678355
- [Background] Galli M, Franchi F, Rollini F, Angiolillo DJ. Role of platelet function and genetic testing in patients undergoing percutaneous coronary intervention. Trends Cardiovasc Med. 2023 Apr;33(3):133-138. doi: 10.1016/j.tcm.2021.12.007. Epub 2021 Dec 20. PMID 34936903
- [Background] Leopold JA, Loscalzo J. Emerging Role of Precision Medicine in Cardiovascular Disease. Circ Res. 2018 Apr 27;122(9):1302-1315. doi: 10.1161/CIRCRESAHA.117.310782. PMID 29700074
- [Background] Claassens DMF, Vos GJA, Bergmeijer TO, Hermanides RS, van 't Hof AWJ, van der Harst P, Barbato E, Morisco C, Tjon Joe Gin RM, Asselbergs FW, Mosterd A, Herrman JR, Dewilde WJM, Janssen PWA, Kelder JC, Postma MJ, de Boer A, Boersma C, Deneer VHM, Ten Berg JM. A Genotype-Guided Strategy for Oral P2Y12 Inhibitors in Primary PCI. N Engl J Med. 2019 Oct 24;381(17):1621-1631. doi: 10.1056/NEJMoa1907096. Epub 2019 Sep 3. PMID 31479209
- [Background] Vyas A, Bash LD, Patel MD, Simpson RJ Jr. Changes in Treatment Patterns and Incremental Health Care Utilization Due to P2Y12-Associated Complications in Patients with Acute Coronary Syndrome. J Manag Care Spec Pharm. 2017 Sep;23(9):947-956. doi: 10.18553/jmcp.2017.23.9.947. PMID 28854078
- [Background] Johnson SG, Gruntowicz D, Chua T, Morlock RJ. Financial Analysis of CYP2C19 Genotyping in Patients Receiving Dual Antiplatelet Therapy Following Acute Coronary Syndrome and Percutaneous Coronary Intervention. J Manag Care Spec Pharm. 2015 Jul;21(7):552-7. doi: 10.18553/jmcp.2015.21.7.552. PMID 26108379
- [Background] Madan M, Abbott JD, Lennon R, So DYF, MacDougall AM, McLaughlin MA, Murthy V, Saw J, Rihal C, Farkouh ME, Pereira NL, Goodman SG; TAILOR-PCI Investigators *. Sex-Specific Differences in Clinical Outcomes After Percutaneous Coronary Intervention: Insights from the TAILOR-PCI Trial. J Am Heart Assoc. 2022 Jun 21;11(12):e024709. doi: 10.1161/JAHA.121.024709. Epub 2022 Jun 14. PMID 35699175
- [Background] Nazir S, Ahuja KR, Virk HUH, Elzanaty A, Waheed TA, Changal KH, Wohlfarth K, Lakhter V, Grande RD, Eltahawy EA. A meta-analysis of efficacy and safety of genotype-guided versus standard of care treatment strategies in selecting antiplatelet therapy in patients with acute coronary syndrome. Catheter Cardiovasc Interv. 2021 Apr 1;97(5):788-794. doi: 10.1002/ccd.28860. Epub 2020 Apr 3. PMID 32243053
- [Background] Nguyen AB, Cavallari LH, Rossi JS, Stouffer GA, Lee CR. Evaluation of race and ethnicity disparities in outcome studies of CYP2C19 genotype-guided antiplatelet therapy. Front Cardiovasc Med. 2022 Aug 23;9:991646. doi: 10.3389/fcvm.2022.991646. eCollection 2022. PMID 36082121
- [Background] Jourdi G, Godier A, Lordkipanidze M, Marquis-Gravel G, Gaussem P. Antiplatelet Therapy for Atherothrombotic Disease in 2022-From Population to Patient-Centered Approaches. Front Cardiovasc Med. 2022 Jan 28;9:805525. doi: 10.3389/fcvm.2022.805525. eCollection 2022. PMID 35155631
- [Background] Urban P, Mehran R, Colleran R, Angiolillo DJ, Byrne RA, Capodanno D, Cuisset T, Cutlip D, Eerdmans P, Eikelboom J, Farb A, Gibson CM, Gregson J, Haude M, James SK, Kim HS, Kimura T, Konishi A, Laschinger J, Leon MB, Magee PFA, Mitsutake Y, Mylotte D, Pocock S, Price MJ, Rao SV, Spitzer E, Stockbridge N, Valgimigli M, Varenne O, Windhoevel U, Yeh RW, Krucoff MW, Morice MC. Defining high bleeding risk in patients undergoing percutaneous coronary intervention: a consensus document from the Academic Research Consortium for High Bleeding Risk. Eur Heart J. 2019 Aug 14;40(31):2632-2653. doi: 10.1093/eurheartj/ehz372. PMID 31116395
- [Background] Palmerini T, Della Riva D, Benedetto U, Bacchi Reggiani L, Feres F, Abizaid A, Gilard M, Morice MC, Valgimigli M, Hong MK, Kim BK, Jang Y, Kim HS, Park KW, Colombo A, Chieffo A, Sangiorgi D, Biondi-Zoccai G, Genereux P, Angelini GD, Pufulete M, White J, Bhatt DL, Stone GW. Three, six, or twelve months of dual antiplatelet therapy after DES implantation in patients with or without acute coronary syndromes: an individual patient data pairwise and network meta-analysis of six randomized trials and 11 473 patients. Eur Heart J. 2017 Apr 7;38(14):1034-1043. doi: 10.1093/eurheartj/ehw627. PMID 28110296
- [Background] Aradi D, Storey RF, Komocsi A, Trenk D, Gulba D, Kiss RG, Husted S, Bonello L, Sibbing D, Collet JP, Huber K; Working Group on Thrombosis of the European Society of Cardiology. Expert position paper on the role of platelet function testing in patients undergoing percutaneous coronary intervention. Eur Heart J. 2014 Jan;35(4):209-15. doi: 10.1093/eurheartj/eht375. Epub 2013 Sep 25. No abstract available. PMID 24067509
- [Background] Capodanno D, Angiolillo DJ. Personalised antiplatelet therapies for coronary artery disease: what the future holds. Eur Heart J. 2023 Aug 22;44(32):3059-3072. doi: 10.1093/eurheartj/ehad362. PMID 37345589
- [Background] van der Sangen NMR, Rozemeijer R, Chan Pin Yin DRPP, Valgimigli M, Windecker S, James SK, Buccheri S, Ten Berg JM, Henriques JPS, Voskuil M, Kikkert WJ. Patient-tailored antithrombotic therapy following percutaneous coronary intervention. Eur Heart J. 2021 Mar 7;42(10):1038-1046. doi: 10.1093/eurheartj/ehaa1097. PMID 33515031
- [Background] Cavallari LH, Beitelshees AL, Blake KV, Dressler LG, Duarte JD, Elsey A, Eichmeyer JN, Empey PE, Franciosi JP, Hicks JK, Holmes AM, Jeng L, Lee CR, Lima JJ, Limdi NA, Modlin J, Obeng AO, Petry N, Pratt VM, Skaar TC, Tuteja S, Voora D, Wagner M, Weitzel KW, Wilke RA, Peterson JF, Johnson JA. The IGNITE Pharmacogenetics Working Group: An Opportunity for Building Evidence with Pharmacogenetic Implementation in a Real-World Setting. Clin Transl Sci. 2017 May;10(3):143-146. doi: 10.1111/cts.12456. Epub 2017 Mar 14. No abstract available. PMID 28294551
- [Background] El Rouby N, Alrwisan A, Langaee T, Lipori G, Angiolillo DJ, Franchi F, Riva A, Elsey A, Johnson JA, Cavallari LH, Winterstein AG. Clinical Utility of Pharmacogene Panel-Based Testing in Patients Undergoing Percutaneous Coronary Intervention. Clin Transl Sci. 2020 May;13(3):473-481. doi: 10.1111/cts.12729. Epub 2020 Jan 16. PMID 31758664
- [Background] Davis BH, DeFrank G, Limdi NA, Harada S. Validation of the Spartan RXCYP2C19 Genotyping Assay Utilizing Blood Samples. Clin Transl Sci. 2020 Mar;13(2):260-264. doi: 10.1111/cts.12714. Epub 2019 Nov 29. PMID 31664775
- [Background] Lee CR, Sriramoju VB, Cervantes A, Howell LA, Varunok N, Madan S, Hamrick K, Polasek MJ, Lee JA, Clarke M, Cicci JD, Weck KE, Stouffer GA. Clinical Outcomes and Sustainability of Using CYP2C19 Genotype-Guided Antiplatelet Therapy After Percutaneous Coronary Intervention. Circ Genom Precis Med. 2018 Apr;11(4):e002069. doi: 10.1161/CIRCGEN.117.002069. PMID 29615454
- [Background] Zhang H, Xiang Q, Liu Z, Mu G, Xie Q, Zhou S, Ma L, Wang Z, Hu K, Wang Z, Cui Y. Genotype-guided antiplatelet treatment versus conventional therapy: A systematic review and meta-analysis. Br J Clin Pharmacol. 2021 May;87(5):2199-2215. doi: 10.1111/bcp.14637. Epub 2020 Dec 29. PMID 33140858
- [Background] Pilling LC, Turkmen D, Fullalove H, Atkins JL, Delgado J, Kuo CL, Kuchel GA, Ferrucci L, Bowden J, Masoli JAH, Melzer D. Analysis of CYP2C19 genetic variants with ischaemic events in UK patients prescribed clopidogrel in primary care: a retrospective cohort study. BMJ Open. 2021 Dec 13;11(12):e053905. doi: 10.1136/bmjopen-2021-053905. PMID 34903548
- [Background] Gower MN, Ratner LR, Williams AK, Rossi JS, Stouffer GA, Lee CR. Clinical Utility of CYP2C19 Genotype-Guided Antiplatelet Therapy in Patients at Risk of Adverse Cardiovascular and Cerebrovascular Events: A Review of Emerging Evidence. Pharmgenomics Pers Med. 2020 Jul 27;13:239-252. doi: 10.2147/PGPM.S231475. eCollection 2020. PMID 32821149
- [Background] Notarangelo FM, Maglietta G, Bevilacqua P, Cereda M, Merlini PA, Villani GQ, Moruzzi P, Patrizi G, Malagoli Tagliazucchi G, Crocamo A, Guidorossi A, Pigazzani F, Nicosia E, Paoli G, Bianchessi M, Comelli MA, Caminiti C, Ardissino D. Pharmacogenomic Approach to Selecting Antiplatelet Therapy in Patients With Acute Coronary Syndromes: The PHARMCLO Trial. J Am Coll Cardiol. 2018 May 1;71(17):1869-1877. doi: 10.1016/j.jacc.2018.02.029. Epub 2018 Mar 11. PMID 29540324
- [Background] Cavallari LH, Lee CR, Beitelshees AL, Cooper-DeHoff RM, Duarte JD, Voora D, Kimmel SE, McDonough CW, Gong Y, Dave CV, Pratt VM, Alestock TD, Anderson RD, Alsip J, Ardati AK, Brott BC, Brown L, Chumnumwat S, Clare-Salzler MJ, Coons JC, Denny JC, Dillon C, Elsey AR, Hamadeh IS, Harada S, Hillegass WB, Hines L, Horenstein RB, Howell LA, Jeng LJB, Kelemen MD, Lee YM, Magvanjav O, Montasser M, Nelson DR, Nutescu EA, Nwaba DC, Pakyz RE, Palmer K, Peterson JF, Pollin TI, Quinn AH, Robinson SW, Schub J, Skaar TC, Smith DM, Sriramoju VB, Starostik P, Stys TP, Stevenson JM, Varunok N, Vesely MR, Wake DT, Weck KE, Weitzel KW, Wilke RA, Willig J, Zhao RY, Kreutz RP, Stouffer GA, Empey PE, Limdi NA, Shuldiner AR, Winterstein AG, Johnson JA; IGNITE Network. Multisite Investigation of Outcomes With Implementation of CYP2C19 Genotype-Guided Antiplatelet Therapy After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2018 Jan 22;11(2):181-191. doi: 10.1016/j.jcin.2017.07.022. Epub 2017 Nov 1. PMID 29102571
- [Background] AlMukdad S, Elewa H, Al-Badriyeh D. Economic Evaluations of CYP2C19 Genotype-Guided Antiplatelet Therapy Compared to the Universal Use of Antiplatelets in Patients With Acute Coronary Syndrome: A Systematic Review. J Cardiovasc Pharmacol Ther. 2020 May;25(3):201-211. doi: 10.1177/1074248420902298. Epub 2020 Feb 6. PMID 32027168
- [Background] Tang B, Wang X, Wang X, Liu L, Ma Z. Genotype-Guided Antiplatelet Therapy Versus Standard Therapy for Patients with Coronary Artery Disease: An Updated Systematic Review and Meta-Analysis. J Pharm Pharm Sci. 2022;25:9-23. doi: 10.18433/jpps32140. PMID 34995471
- [Background] Leucht S, Helfer B, Gartlehner G, Davis JM. How effective are common medications: a perspective based on meta-analyses of major drugs. BMC Med. 2015 Oct 2;13:253. doi: 10.1186/s12916-015-0494-1. PMID 26431961
- [Background] Yamani N, Unzek S, Mankani MH, Almas T, Musheer A, Qamar H, Farooq S, Shahnawaz W, Fatima K, Figueredo V, Mookadam F. Does individualized guided selection of antiplatelet therapy improve outcomes after percutaneous coronary intervention? A systematic review and meta-analysis. Ann Med Surg (Lond). 2022 Jun 18;79:103964. doi: 10.1016/j.amsu.2022.103964. eCollection 2022 Jul. PMID 35860051
- [Background] Lee SH, Jeong YH, Hong D, Choi KH, Lee JM, Park TK, Yang JH, Hahn JY, Choi SH, Gwon HC, Jeong MH, Kim BK, Joo HJ, Chang K, Park Y, Ahn SG, Suh JW, Lee SY, Cho JR, Her AY, Kim HS, Kim MH, Lim DS, Shin ES, Song YB; PTRG-DES Registry Investigators. Clinical Impact of CYP2C19 Genotype on Clopidogrel-Based Antiplatelet Therapy After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2023 Apr 10;16(7):829-843. doi: 10.1016/j.jcin.2023.01.363. Epub 2023 Mar 8. PMID 37045504
- [Background] Ingraham BS, Farkouh ME, Lennon RJ, So D, Goodman SG, Geller N, Bae JH, Jeong MH, Baudhuin LM, Mathew V, Bell MR, Lerman A, Fu YP, Hasan A, Iturriaga E, Tanguay JF, Welsh RC, Rosenberg Y, Bailey K, Rihal C, Pereira NL. Genetic-Guided Oral P2Y12 Inhibitor Selection and Cumulative Ischemic Events After Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2023 Apr 10;16(7):816-825. doi: 10.1016/j.jcin.2023.01.356. PMID 37045502
- [Background] Stys TP, Gedela M, Gowda SN, Bares V, Fanta L, Petrasko M, Hajek C, Larson E, Stys AT. CYP2C19 genotype-directed P2Y12 inhibitor antiplatelet therapy normalizes risk for major adverse cardiovascular events after percutaneous coronary intervention. Indian Heart J. 2021 May-Jun;73(3):281-288. doi: 10.1016/j.ihj.2021.03.004. Epub 2021 Mar 17. PMID 34154743
- [Background] Pereira NL, Rihal CS, So DYF, Rosenberg Y, Lennon RJ, Mathew V, Goodman SG, Weinshilboum RM, Wang L, Baudhuin LM, Lerman A, Hasan A, Iturriaga E, Fu YP, Geller N, Bailey K, Farkouh ME. Clopidogrel Pharmacogenetics. Circ Cardiovasc Interv. 2019 Apr;12(4):e007811. doi: 10.1161/CIRCINTERVENTIONS.119.007811. PMID 30998396
- [Background] Tuteja S, Glick H, Matthai W, Nachamkin I, Nathan A, Monono K, Carcuffe C, Maslowski K, Chang G, Kobayashi T, Anwaruddin S, Hirshfeld J, Wilensky RL, Herrmann HC, Kolansky DM, Rader DJ, Giri J. Prospective CYP2C19 Genotyping to Guide Antiplatelet Therapy Following Percutaneous Coronary Intervention: A Pragmatic Randomized Clinical Trial. Circ Genom Precis Med. 2020 Feb;13(1):e002640. doi: 10.1161/CIRCGEN.119.002640. Epub 2020 Jan 12. PMID 31928229
- [Background] Lee CR, Luzum JA, Sangkuhl K, Gammal RS, Sabatine MS, Stein CM, Kisor DF, Limdi NA, Lee YM, Scott SA, Hulot JS, Roden DM, Gaedigk A, Caudle KE, Klein TE, Johnson JA, Shuldiner AR. Clinical Pharmacogenetics Implementation Consortium Guideline for CYP2C19 Genotype and Clopidogrel Therapy: 2022 Update. Clin Pharmacol Ther. 2022 Nov;112(5):959-967. doi: 10.1002/cpt.2526. Epub 2022 Feb 8. PMID 35034351
- [Background] Abdullah-Koolmees H, van Keulen AM, Nijenhuis M, Deneer VHM. Pharmacogenetics Guidelines: Overview and Comparison of the DPWG, CPIC, CPNDS, and RNPGx Guidelines. Front Pharmacol. 2021 Jan 25;11:595219. doi: 10.3389/fphar.2020.595219. eCollection 2020. PMID 33568995
- [Background] Dayoub EJ, Seigerman M, Tuteja S, Kobayashi T, Kolansky DM, Giri J, Groeneveld PW. Trends in Platelet Adenosine Diphosphate P2Y12 Receptor Inhibitor Use and Adherence Among Antiplatelet-Naive Patients After Percutaneous Coronary Intervention, 2008-2016. JAMA Intern Med. 2018 Jul 1;178(7):943-950. doi: 10.1001/jamainternmed.2018.0783. PMID 29799992
- [Background] Parcha V, Heindl BF, Li P, Kalra R, Limdi NA, Pereira NL, Arora G, Arora P. Genotype-Guided P2Y12 Inhibitor Therapy After Percutaneous Coronary Intervention: A Bayesian Analysis. Circ Genom Precis Med. 2021 Dec;14(6):e003353. doi: 10.1161/CIRCGEN.121.003353. Epub 2021 Oct 21. PMID 34670396
- [Background] Pereira NL, Farkouh ME, So D, Lennon R, Geller N, Mathew V, Bell M, Bae JH, Jeong MH, Chavez I, Gordon P, Abbott JD, Cagin C, Baudhuin L, Fu YP, Goodman SG, Hasan A, Iturriaga E, Lerman A, Sidhu M, Tanguay JF, Wang L, Weinshilboum R, Welsh R, Rosenberg Y, Bailey K, Rihal C. Effect of Genotype-Guided Oral P2Y12 Inhibitor Selection vs Conventional Clopidogrel Therapy on Ischemic Outcomes After Percutaneous Coronary Intervention: The TAILOR-PCI Randomized Clinical Trial. JAMA. 2020 Aug 25;324(8):761-771. doi: 10.1001/jama.2020.12443. PMID 32840598
- [Background] Chanfreau-Coffinier C, Friede KA, Plomondon ME, Lee KM, Lu Z, Lynch JA, DuVall SL, Vassy JL, Waldo SW, Cleator JH, Maddox TM, Rader DJ, Assimes TL, Damrauer SM, Tsao PS, Chang KM, Voora D, Giri J, Tuteja S. CYP2C19 Polymorphisms and Clinical Outcomes Following Percutaneous Coronary Intervention (PCI) in the Million Veterans Program. medRxiv [Preprint]. 2023 Oct 26:2023.10.25.23297578. doi: 10.1101/2023.10.25.23297578. PMID 37961335
- [Background] Martin J, Williams AK, Klein MD, Sriramoju VB, Madan S, Rossi JS, Clarke M, Cicci JD, Cavallari LH, Weck KE, Stouffer GA, Lee CR. Frequency and clinical outcomes of CYP2C19 genotype-guided escalation and de-escalation of antiplatelet therapy in a real-world clinical setting. Genet Med. 2020 Jan;22(1):160-169. doi: 10.1038/s41436-019-0611-1. Epub 2019 Jul 18. PMID 31316169
- [Background] Sibbing D, Aradi D, Alexopoulos D, Ten Berg J, Bhatt DL, Bonello L, Collet JP, Cuisset T, Franchi F, Gross L, Gurbel P, Jeong YH, Mehran R, Moliterno DJ, Neumann FJ, Pereira NL, Price MJ, Sabatine MS, So DYF, Stone GW, Storey RF, Tantry U, Trenk D, Valgimigli M, Waksman R, Angiolillo DJ. Updated Expert Consensus Statement on Platelet Function and Genetic Testing for Guiding P2Y12 Receptor Inhibitor Treatment in Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2019 Aug 26;12(16):1521-1537. doi: 10.1016/j.jcin.2019.03.034. Epub 2019 Jun 12. PMID 31202949
- [Background] Capodanno D, Angiolillo DJ, Lennon RJ, Goodman SG, Kim SW, O'Cochlain F, So DY, Sweeney J, Rihal CS, Farkouh M, Pereira NL. ABCD-GENE Score and Clinical Outcomes Following Percutaneous Coronary Intervention: Insights from the TAILOR-PCI Trial. J Am Heart Assoc. 2022 Feb 15;11(4):e024156. doi: 10.1161/JAHA.121.024156. Epub 2022 Feb 8. PMID 35132875
- [Background] Al-Abcha A, Radwan Y, Blais D, Mazzaferri EL Jr, Boudoulas KD, Essa EM, Gumina RJ. Genotype-Guided Use of P2Y12 Inhibitors: A Review of Current State of the Art. Front Cardiovasc Med. 2022 Mar 23;9:850028. doi: 10.3389/fcvm.2022.850028. eCollection 2022. PMID 35402528
- [Background] Dannenberg L, Afzal S, Czychy N, M'Pembele R, Zako S, Helten C, Mourikis P, Zikeli D, Ahlbrecht S, Trojovsky K, Benkhoff M, Barcik M, Wolff G, Zeus T, Kelm M, Polzin A. Risk prediction of bleeding and MACCE by PRECISE-DAPT score post-PCI. Int J Cardiol Heart Vasc. 2021 Mar 13;33:100750. doi: 10.1016/j.ijcha.2021.100750. eCollection 2021 Apr. PMID 33763519
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC Jr. 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention, 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery, 2012 ACC/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the Diagnosis and Management of Patients With Stable Ischemic Heart Disease, 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction, 2014 AHA/ACC Guideline for the Management of Patients With Non-ST-Elevation Acute Coronary Syndromes, and 2014 ACC/AHA Guideline on Perioperative Cardiovascular Evaluation and Management of Patients Undergoing Noncardiac Surgery. Circulation. 2016 Sep 6;134(10):e123-55. doi: 10.1161/CIR.0000000000000404. Epub 2016 Mar 29. No abstract available. PMID 27026020
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Background] Luengo-Fernandez R, Walli-Attaei M, Gray A, Torbica A, Maggioni AP, Huculeci R, Bairami F, Aboyans V, Timmis AD, Vardas P, Leal J. Economic burden of cardiovascular diseases in the European Union: a population-based cost study. Eur Heart J. 2023 Dec 1;44(45):4752-4767. doi: 10.1093/eurheartj/ehad583. PMID 37632363
- [Background] Crea F, Libby P. Acute Coronary Syndromes: The Way Forward From Mechanisms to Precision Treatment. Circulation. 2017 Sep 19;136(12):1155-1166. doi: 10.1161/CIRCULATIONAHA.117.029870. PMID 28923905
- See also: Clopidogrel, Drug Usage Statistics, United States, 2013 - 2022 — https://clincalc.com/DrugStats/Drugs/Clopidogrel
- See also: CPIC® Guideline for Clopidogrel and CYP2C19 — https://cpicpgx.org/guidelines/guideline-for-clopidogrel-and-cyp2c19/
- See also: PharmGKB Clinical Annotations of Clopidogrel, information about variant-drug pairs based primarily on variant annotations and incorporating variant-specific prescribing guidance from clinical guidelines and FDA-approved drug labels, when available. — https://www.pharmgkb.org/chemical/PA449053/clinicalAnnotation
- See also: Dean L, Kane M. Clopidogrel Therapy and CYP2C19 Genotype. 2012 Mar 8 [Updated 2022 Dec 1]. In: Pratt VM, Scott SA, Pirmohamed M, et al., editors. Medical Genetics Summaries [Internet]. Bethesda (MD): National Center for Biotechnology Information (US); 20 — https://www.ncbi.nlm.nih.gov/books/NBK84114/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study investigating CYP2C19 genotype-guided clopidogrel treatment models was conducted by Vistamedi Ltd. (Tbilisi, Georgia) collecting data from out-patient and hospital health care facilities of four clinical cardiology centers in Tbilisi, Georgia.
  The active recruitment process started after obtaining Institutional Review Boars (IRB) approval of the study protocol and continued for 12 months.
Pre-assignment Details: In total, 330 study participants were screened for participation, and 283 who met the study eligibility criteria and signed informed consent forms for study participation were recruited.
Period: Overall Study
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Started | 157 | 43 | 83
Completed | 142 | 38 | 70
Not Completed | 15 | 5 | 13
Not completed — Withdrawal by Subject | 4 | 4 | 4
Not completed — Non-compliance to Treatment | 4 | 1 | 6
Not completed — Lost to Follow-up | 3 | 0 | 2
Not completed — Physician Decision | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Study participants of both sexes aged 35-79 years old, diagnosed with chronic coronary artery disease who had undergone elective PCI and required P2Y12 inhibitor antiplatelet treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel | Total
Number analyzed (Participants) | 157 | 43 | 83 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The mean age of study arm participants is given for overall and sex-specific groups
  years
    mean age of overall study participants | 63.91 (9.03) | 66.35 (7.34) | 63.49 (9.96) | 64.16 (9.10)
    mean age of female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    mean age of female study participants | 68.73 (7.15) | 69.25 (6.96) | 67.80 (8.05) | 68.57 (7.33)
    mean age of male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    mean age of male study participants | 61.24 (8.88) | 63.83 (6.84) | 61.06 (10.18) | 61.52 (9.06)
Age, Customized [Count of Participants; unit: Participants]
  Age ranges of study participants: 35-49 years old | 13 | 0 | 8 | 21
  Age ranges of study participants: 50-64 years old | 62 | 17 | 33 | 112
  Age ranges of study participants: 65-79 years old | 82 | 26 | 42 | 150
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 20 | 30 | 106
  Male | 101 | 23 | 53 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 157 | 43 | 83 | 283
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Georgia | 157 | 43 | 83 | 283
Smoking status of study participants [Count of Participants; unit: Participants] — Smoking status measured as number and percentage of Current Smokers, Former Smokers and Never Smokers among study participants Population: Smoking status patterns among overall, sex-specific and age-specific study participants groups
  Participants
    Overall study participants: Current Smoker | 58 | 14 | 50 | 122
    Overall study participants: Former Smoker | 57 | 16 | 14 | 87
    Overall study participants: Never Smoker | 42 | 13 | 19 | 74
    Female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    Female study participants: Current Smoker | 7 | 1 | 7 | 15
    Female study participants: Former Smoker | 12 | 6 | 5 | 23
    Female study participants: Never Smoker | 37 | 13 | 18 | 68
    Male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    Male study participants: Current Smoker | 51 | 13 | 43 | 107
    Male study participants: Former Smoker | 45 | 10 | 9 | 64
    Male study participants: Never Smoker | 5 | 0 | 1 | 6
    35-49 years old study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    35-49 years old study participants: Current Smoker | 8 | 0 | 7 | 15
    35-49 years old study participants: Former Smoker | 4 | 0 | 1 | 5
    35-49 years old study participants: Never Smoker | 1 | 0 | 0 | 1
    50-64 years old study participants: number analyzed (Participants) | 62 | 17 | 33 | 112
    50-64 years old study participants: Current Smoker | 34 | 8 | 29 | 71
    50-64 years old study participants: Former Smoker | 20 | 7 | 3 | 30
    50-64 years old study participants: Never Smoker | 8 | 2 | 1 | 11
    65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    65-79 years old study participants: Current Smoker | 16 | 6 | 14 | 36
    65-79 years old study participants: Former Smoker | 33 | 9 | 10 | 52
    65-79 years old study participants: Never Smoker | 33 | 11 | 18 | 62
Obesity among study participants [Count of Participants; unit: Participants] — Number and percentage of study participants with obesity (BMI =>30kg/m^2 but <=40kg/m^2) Population: Number and percentage of obese study participants in the overall, sex- and age-specific groups
  Participants
    Overall study participants | 91 | 21 | 48 | 160
    Female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    Female study participants | 31 | 10 | 22 | 63
    Male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    Male study participants | 60 | 11 | 26 | 97
    35-49 years study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    35-49 years study participants | 7 | 0 | 6 | 13
    50-64 years old study participants: number analyzed (Participants) | 62 | 17 | 33 | 112
    50-64 years old study participants | 53 | 8 | 17 | 78
    65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    65-79 years old study participants | 41 | 13 | 25 | 79
Body Mass Index (BMI) of study participants [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) of study participants measured as Body Weight/Body Height^2 (kg/m^2) Population: The mean BMI (kg/m^2) of overall, sex- and age-specific group study participants
  kg/m^2
    Overall study participants | 30.5 (4.32) | 30.5 (4.67) | 31.0 (3.65) | 30.6 (4.18)
    Female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    Female study participants | 30.2 (4.62) | 30.5 (4.88) | 31.7 (3.12) | 30.7 (4.31)
    Male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    Male study participants | 30.6 (4.17) | 30.5 (4.58) | 30.57 (3.89) | 30.6 (4.12)
    35-49 years old study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    35-49 years old study participants | 30.2 (4.69) |  | 31.6 (3.70) | 30.7 (4.30)
    50-64 years old study participants: number analyzed (Participants) | 62 | 17 | 33 | 112
    50-64 years old study participants | 31.3 (4.00) | 30.8 (5.20) | 30.6 (2.90) | 31.00 (3.90)
    65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    65-79 years old study participants | 29.9 (4.46) | 30.3 (4.38) | 31.1 (4.18) | 30.3 (4.37)
Blood Pressure control [Count of Participants; unit: Participants] — Blood pressure (BP) controlling status assessed as controlled (SBP<140mmHg and DBP<90mmHg) or uncontrolled (SBP>/=140mmHg and/or DBP>/=90mmHg) at the time of study enrollment Population: Number and percentage of study participants with controlled and uncontrolled blood pressure in the overall, and sex- and age-specific groups
  Participants
    Overall study participants: with Controlled BP | 89 | 28 | 21 | 138
    Overall study participants: with Uncontrolled BP | 68 | 15 | 62 | 145
    Female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    Female study participants: with Controlled BP | 31 | 13 | 7 | 51
    Female study participants: with Uncontrolled BP | 25 | 7 | 23 | 55
    Male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    Male study participants: with Controlled BP | 58 | 15 | 14 | 87
    Male study participants: with Uncontrolled BP | 43 | 8 | 39 | 90
    35-49 years old study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    35-49 years old study participants: with Controlled BP | 8 | 0 | 5 | 13
    35-49 years old study participants: with Uncontrolled BP | 5 | 0 | 3 | 8
    50-64 years old study participants: number analyzed (Participants) | 62 | 17 | 33 | 112
    50-64 years old study participants: with Controlled BP | 34 | 11 | 8 | 53
    50-64 years old study participants: with Uncontrolled BP | 28 | 6 | 25 | 59
    65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    65-79 years old study participants: with Controlled BP | 47 | 17 | 8 | 72
    65-79 years old study participants: with Uncontrolled BP | 35 | 9 | 34 | 78
BP measurement results of study participants [Mean (Standard Deviation); unit: mmHg] — SBP and DBP measurement results (mmHg) of study participants at the time of study enrollment Population: The mean SBP and DBP (mmHg) of study participants overall, and by sex- and age-specific groups
  mmHg
    SBP of overall study participants | 138.1 (21.44) | 134.1 (19.57) | 149.0 (16.27) | 140.7 (20.47)
    DBP of overall study participants | 82.4 (12.19) | 79.6 (12.45) | 89.3 (10.52) | 84.0 (12.25)
    SBP of female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    SBP of female study participants | 139.1 (22.64) | 135.9 (20.27) | 150.1 (17.84) | 141.6 (21.47)
    DBP of female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    DBP of female study participants | 82.7 (11.75) | 78.7 (12.89) | 88.6 (10.20) | 83.6 (11.97)
    SBP of male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    SBP of male study participants | 137.5 (20.83) | 132.5 (19.26) | 148.3 (15.45) | 140.1 (19.88)
    DBP of male study participant: number analyzed (Participants) | 101 | 23 | 53 | 177
    DBP of male study participant | 82.2 (12.47) | 80.4 (12.28) | 89.7 (10.77) | 84.2 (12.44)
    SBP of 35-49 years old study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    SBP of 35-49 years old study participants | 129.5 (12.61) |  | 135.0 (15.34) | 131.6 (13.62)
    DBP of 35-49 years old study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    DBP of 35-49 years old study participants | 83.8 (10.34) |  | 83.5 (12.50) | 83.7 (10.90)
    SBP of 50-64 years old study participant: number analyzed (Participants) | 62 | 17 | 33 | 112
    SBP of 50-64 years old study participant | 139.9 (21.55) | 133.7 (20.01) | 150.4 (16.16) | 142.1 (20.55)
    DBP of 50-64 years old study participants: number analyzed (Participants) | 62 | 17 | 33 | 112
    DBP of 50-64 years old study participants | 83.3 (13.51) | 80.5 (12.97) | 91.3 (10.74) | 85.2 (13.22)
    SBP of 65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    SBP of 65-79 years old study participants | 138.0 (22.31) | 134.3 (19.68) | 150.5 (15.59) | 140.8 (20.98)
    DBP of 65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    DBP of 65-79 years old study participants | 81.5 (11.45) | 79.1 (12.32) | 88.8 (9.71) | 83.1 (11.67)
Type 2 Diabetes Mellitus [Count of Participants; unit: Participants] — Type 2 Diabetes Mellitus (T2DM) control status of study participant measured as Uncontrolled (diagnosed T2DM and glycated hemoglobin (HbA1c) is >/=6.2%), Controlled (diagnosed T2DM and HbA1c is <6.2%) and No T2DM (not diagnosed T2DM and HbA1c is <6.2%) Population: Number and percentage of study participants with Uncontrolled, Controlled and No T2DM in overall, by sex- and age-specific arms at the time of enrollment
  Participants
    Overall study participants: Uncontrolled T2DM | 59 | 16 | 40 | 115
    Overall study participants: Controlled T2DM | 30 | 8 | 3 | 41
    Overall study participants: No T2DM | 68 | 19 | 40 | 127
    Female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    Female study participants: Uncontrolled T2DM | 16 | 10 | 16 | 42
    Female study participants: Controlled T2DM | 15 | 4 | 1 | 20
    Female study participants: No T2DM | 25 | 6 | 13 | 44
    Male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    Male study participants: Uncontrolled T2DM | 43 | 6 | 24 | 73
    Male study participants: Controlled T2DM | 15 | 4 | 2 | 21
    Male study participants: No T2DM | 43 | 13 | 27 | 83
    35-49 years old study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    35-49 years old study participants: Uncontrolled T2DM | 6 | 0 | 2 | 8
    35-49 years old study participants: Controlled T2DM | 0 | 0 | 1 | 1
    35-49 years old study participants: No T2DM | 7 | 0 | 5 | 12
    40-64 years old study participants: number analyzed (Participants) | 62 | 17 | 33 | 112
    40-64 years old study participants: Uncontrolled T2DM | 26 | 5 | 15 | 46
    40-64 years old study participants: Controlled T2DM | 12 | 1 | 2 | 15
    40-64 years old study participants: No T2DM | 24 | 11 | 16 | 51
    65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    65-79 years old study participants: Uncontrolled T2DM | 27 | 11 | 23 | 61
    65-79 years old study participants: Controlled T2DM | 18 | 7 | 0 | 25
    65-79 years old study participants: No T2DM | 37 | 8 | 19 | 64
Glycated Hemoglobin (HbA1c) Levels [Mean (Standard Deviation); unit: percentage (%) of glycated hemoglobin] — HbA1c (%) measurement results of study participants Population: Mean HbA1c measurement results (in %) of study participants overall, and by sex- and age-specific groups
  percentage (%) of glycated hemoglobin
    Overall study participants | 6.3 (0.94) | 6.3 (1.01) | 6.5 (1.13) | 6.4 (1.01)
    Female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    Female study participants | 6.1 (0.78) | 6.7 (1.12) | 6.6 (1.23) | 6.4 (1.02)
    Male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    Male study participants | 6.5 (1.01) | 6.0 (0.78) | 6.5 (1.08) | 6.4 (0.95)
    35-49 years old study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    35-49 years old study participants | 6.5 (1.07) |  | 6.2 (1.11) | 6.4 (1.07)
    50-64 years old study participants: number analyzed (Participants) | 62 | 17 | 33 | 112
    50-64 years old study participants | 6.4 (1.05) | 6.1 (0.97) | 6.5 (1.13) | 6.4 (1.06)
    65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    65-79 years old study participants | 6.2 (0.83) | 6.5 (1.01) | 6.7 (1.15) | 6.4 (0.98)
Low Density Lipoprotein Cholesterol (LDL-C) Controlling Status [Count of Participants; unit: Participants] — Serum Low Density Lipoprotein Cholesterol (LDL) control status measured as Controlled (LDL-C <55mg/dl ) or Uncontrolled (LDL-C >/=55mg/dl) Population: Number and percentage of study participants with uncontrolled and controlled LDL-C levels in the overall, and by sex- and age-specific groups
  Participants
    Overall study participants: Uncontrolled LDL-C Level | 92 | 18 | 71 | 181
    Overall study participants: Controlled LDL-C Level | 65 | 25 | 12 | 102
    Female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    Female study participants: Uncontrolled LDL-C Level | 32 | 7 | 28 | 67
    Female study participants: Controlled LDL-C Level | 24 | 13 | 2 | 39
    Male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    Male study participants: Uncontrolled LDL-C Level | 60 | 11 | 43 | 114
    Male study participants: Controlled LDL-C Level | 41 | 12 | 10 | 63
    35-49 years old study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    35-49 years old study participants: Uncontrolled LDL-C Level | 9 | 0 | 4 | 13
    35-49 years old study participants: Controlled LDL-C Level | 4 | 0 | 4 | 8
    50-64 years old study participants: number analyzed (Participants) | 62 | 17 | 33 | 112
    50-64 years old study participants: Uncontrolled LDL-C Level | 33 | 5 | 29 | 67
    50-64 years old study participants: Controlled LDL-C Level | 29 | 12 | 4 | 45
    65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    65-79 years old study participants: Uncontrolled LDL-C Level | 50 | 13 | 38 | 101
    65-79 years old study participants: Controlled LDL-C Level | 32 | 13 | 4 | 49
Serum LDL-C measurement results [Mean (Standard Deviation); unit: mg/dl] — The mean serum LDL-C measurement results (in mg/dl) of study participants at the time of enrollment Population: The mean LDL-C level of study participants overall, and by sex- and age-specific groups
  mg/dl
    Overall study participants | 94.6 (51.59) | 77.6 (42.59) | 117.5 (35.56) | 98.7 (47.87)
    Female study participants: number analyzed (Participants) | 56 | 20 | 30 | 106
    Female study participants | 91.8 (48.85) | 73.2 (39.87) | 119.9 (25.49) | 96.2 (44.59)
    Male study participants: number analyzed (Participants) | 101 | 23 | 53 | 177
    Male study participants | 96.1 (53.23) | 81.4 (45.35) | 116.1 (40.33) | 100.2 (49.80)
    35-49 years old study participants: number analyzed (Participants) | 13 | 0 | 8 | 21
    35-49 years old study participants | 99.5 (57.12) |  | 95.6 (55.01) | 98.0 (55.03)
    50-64 years old study participants: number analyzed (Participants) | 62 | 17 | 33 | 112
    50-64 years old study participants | 95.0 (53.93) | 70.3 (46.2) | 118.3 (34.45) | 98.1 (49.93)
    65-79 years old study participants: number analyzed (Participants) | 82 | 26 | 42 | 150
    65-79 years old study participants | 93.5 (49.47) | 82.4 (40.26) | 121.0 (31.29) | 99.3 (45.54)
Symptom manifestations/conditions prior to index PCI [Count of Participants; unit: Participants] — Any cardiovascular disease/condition present in the past medical history Population: Number and percentage of study participants with angina and other clinical conditions considered as the reason for the most recent PCI
  Participants
    Angina | 107 | 28 | 76 | 211
    No angina | 50 | 15 | 7 | 72
    Heart Failure Event: number analyzed (Participants) | 50 | 15 | 7 | 72
    Heart Failure Event | 22 | 5 | 5 | 32
    Supraventricular Tachycardia: number analyzed (Participants) | 50 | 15 | 7 | 72
    Supraventricular Tachycardia | 5 | 2 | 1 | 8
    Atrial Fibrillation: number analyzed (Participants) | 50 | 15 | 7 | 72
    Atrial Fibrillation | 7 | 2 | 0 | 9
    Premature Ventricular Contraction/Ventricular tachycardia: number analyzed (Participants) | 50 | 15 | 7 | 72
    Premature Ventricular Contraction/Ventricular tachycardia | 1 | 1 | 0 | 2
    Left Bundle Branch Block: number analyzed (Participants) | 50 | 15 | 7 | 72
    Left Bundle Branch Block | 2 | 0 | 0 | 2
    Other non-specific symptoms: number analyzed (Participants) | 50 | 15 | 7 | 72
    Other non-specific symptoms | 13 | 5 | 1 | 19
History of Cardiovascular Morbidity [Count of Participants; unit: Participants] — The number and percentage (%) of study participants with any cardiovascular disease/condition presented in the past medical history
  Participants
    Prior Myocardium Infarction | 83 | 21 | 40 | 144
    Chronic Heart Failure | 50 | 13 | 29 | 92
    Supraventricular tachycardia - paroxysmal | 29 | 6 | 2 | 37
    Supraventricular tachycardia - paroxysmal, recurrent | 6 | 4 | 0 | 10
    Atrial Fibrillation - Paroxysmal | 3 | 1 | 2 | 6
    Atrial Fibrillation - Persistent | 23 | 6 | 5 | 34
    Atrial Fibrillation - Permanent | 5 | 2 | 4 | 11
    Premature Ventricular Contraction | 135 | 35 | 80 | 250
    Ventricular Tachycardia | 25 | 5 | 4 | 34
    Ventricular Fibrillation Event | 8 | 0 | 1 | 9
    Sinus Node Disfunction | 4 | 1 | 1 | 6
    AV Block | 10 | 0 | 3 | 13
    Left Bundle Branch Block | 19 | 4 | 17 | 40
    Bight Bundle Branch Block | 40 | 18 | 23 | 81
Coronary artery bypass grafting [Count of Participants; unit: Participants] — The number and percentage of study participants undergone coronary artery bypass grafting (CABG) in the past medical history
  Participants | 21 | 5 | 7 | 33
Major Coronary Vascular Event [Mean (Standard Deviation); unit: number of events] — The mean number of non-fatal major coronary vascular event assessed as prior myocardium infarction and PCIs underwent in the past medical history
  number of events
    Number of Prior MI events | 0.53 (0.51) | 0.49 (0.51) | 0.55 (0.63) | 0.53 (0.53)
    Number of PCIs | 1.55 (0.58) | 1.56 (0.67) | 1.75 (0.71) | 1.61 (0.64)
Atherosclerotic vascular co-morbid diseases/conditions [Count of Participants; unit: Participants] — Number and percentage of study participants priorly diagnosed atherosclerotic vascular co-morbid diseases/conditions in the past medical history
  Participants
    Peripheral Artery Disease without intravascular intervention | 15 | 7 | 9 | 31
    Peripheral Artery Disease with endarterectomy | 2 | 0 | 1 | 3
    Peripheral Artery Disease with stenting | 6 | 2 | 11 | 19
    Peripheral Artery Disease with endarterectomy and stenting | 3 | 1 | 0 | 4
    Carotid Artery Disease without intravascular intervention | 36 | 9 | 22 | 67
    Carotid Artery Disease with endarterectomy | 4 | 0 | 8 | 12
    Carotid Artery Disease with stenting | 1 | 2 | 0 | 3
    Carotid Artery Disease with endarterectomy and stenting | 2 | 0 | 0 | 2
    Cerebrovascular Disease with minor stroke | 14 | 2 | 0 | 16
    Cerebrovascular Disease with TIA | 51 | 15 | 30 | 96
Other co-morbid diseases/conditions [Count of Participants; unit: Participants] — Number and percentage of study participants priorly diagnosed with other co-morbid diseases/conditions in the past medical history
  Participants
    Chronic Obstructive Pulmonary Disease | 55 | 13 | 26 | 94
    Chronic Kidney Disease | 36 | 8 | 26 | 70
    Peptic Ulcer | 21 | 11 | 12 | 44
    Chronic Gastritis | 59 | 18 | 30 | 107
    GI Bleeding Event | 7 | 2 | 6 | 15
    Cured Cancer | 14 | 5 | 8 | 27
    Thyroid Disease | 25 | 8 | 5 | 38
Coronary Artery Lesion [Mean (Standard Deviation); unit: Coronary artery lesions] — The mean number of any and haemodynamically significant (>50% stenosis in the left main - LM, or ≥70% stenosis in the left anterior descending - LAD, the left circumflex - LCX, and the right coronary - RCA) lesion sites of coronary arteries
  Coronary artery lesions
    Total Number of Coronary Artery Lesion Sites | 4.01 (1.10) | 3.79 (1.13) | 4.17 (1.09) | 4.01 (1.10)
    Number of Haemodynamically Significant Coronary Artery Lesion Sites | 2.53 (1.21) | 2.23 (0.95) | 2.54 (1.10) | 2.49 (1.14)
Intracoronary Stenting History [Mean (Standard Deviation); unit: number of stents] — The number of intracoronary stents ever placed
  number of stents | 2.17 (0.88) | 2.09 (0.72) | 2.33 (0.98) | 2.20 (0.89)
Coronary Artery Anatomy [Count of Participants; unit: Participants] — Number and percentage of study participants with obstructive or non-obstructive lesions of the certain coronary arteries assessed by coronary angiography at the time of index PCI
  Participants
    Left main coronary artery : Obstructive | 5 | 0 | 0 | 5
    Left main coronary artery : Non-obstructive | 6 | 3 | 4 | 13
    Left anterior descending artery : Obstructive | 105 | 30 | 52 | 187
    Left anterior descending artery : Non-obstructive | 15 | 5 | 11 | 31
    1st diagonal branch of the left anterior descending coronary artery : Obstructive | 56 | 12 | 29 | 97
    1st diagonal branch of the left anterior descending coronary artery : Non-obstructive | 30 | 7 | 17 | 54
    2nd diagonal branch of the left anterior descending coronary artery : Obstructive | 4 | 2 | 3 | 9
    2nd diagonal branch of the left anterior descending coronary artery : Non-obstructive | 9 | 2 | 7 | 18
    Left circumflex artery : Obstructive | 104 | 26 | 53 | 183
    Left circumflex artery : Non-obstructive | 26 | 12 | 17 | 55
    1st Marginal arteries : Obstructive | 40 | 9 | 24 | 73
    1st Marginal arteries : Non-obstructive | 39 | 14 | 29 | 82
    2nd Marginal arteries : Obstructive | 1 | 1 | 1 | 3
    2nd Marginal arteries : Non-obstructive | 7 | 0 | 3 | 10
    Right coronary artery : Obstructive | 75 | 20 | 34 | 129
    Right coronary artery : Non-obstructive | 44 | 15 | 25 | 84
    Right marginal branch of right coronary artery : Obstructive | 1 | 0 | 0 | 1
    Right marginal branch of right coronary artery : Non-obstructive | 2 | 1 | 0 | 3
    Posterior descending artery : Obstructive | 12 | 2 | 15 | 29
    Posterior descending artery : Non-obstructive | 13 | 2 | 8 | 23
Echocardiographic Linear Dimensions [Mean (Standard Deviation); unit: millimeter] — Mean linear dimension values of cardiac structural elements measured by echocardiographic imaging
  millimeter
    Left ventricular posterior wall thickness | 11.45 (1.22) | 11.30 (1.01) | 11.54 (1.73) | 11.46 (1.86)
    Interventricular septum thickness | 12.04 (1.33) | 11.88 (1.14) | 12.49 (1.84) | 12.15 (1.49)
    Left ventricular end-diastolic diameter | 49.64 (5.49) | 48.02 (4.07) | 50.41 (4.58) | 49.62 (5.27)
    Left atrium transverse diameter | 42.51 (5.87) | 42.84 (4.07) | 41.36 (5.37) | 42.22 (5.50)
Left Ventricular Volume Index [Mean (Standard Deviation); unit: milliliter per square meter (ml/m^2)] — Left ventricular end-diastolic volume in millilitres measured by the biplane area-length method using 4- and 2-chamber views with two-dimensional echocardiographic imaging and indexed with the patient's body surface area in square meters calculated by the Du Bois formula
  milliliter per square meter (ml/m^2) | 64.87 (20.53) | 60.70 (18.35) | 56.04 (10.58) | 61.64 (18.19)
Left Atrium Volume Index [Mean (Standard Deviation); unit: millilitre per square meter (ml/m^2)] — Left atrium end-systolic volume in millilitres measured by biplane area-length method using 4- and 2-chamber views with two-dimensional echocardiographic assessment and indexed with the patient's body surface area in square meters calculated by the Du Bois formula
  millilitre per square meter (ml/m^2) | 37.45 (5.89) | 36.56 (5.86) | 37.47 (5.41) | 37.32 (5.73)
Left Ventricular Mass Index [Mean (Standard Deviation); unit: gram per square meter (g/m^2)] — Left ventricular myocardium mass in grams calculated by Deverioux regression model formula using linear sizes of left ventricular posterior wall thickness, interventricular septum thickness and end-diastolic cavity diameter in centimeters with retraction of left ventricular cavity volume from volume enclosed by epicardium to obtain the net myocardium volume in millilitres, than multiplicated by the myocardium density measured in grams per millilitre and indexed with the patient's body surface area in square meters calculated by the Du Bois formula
  gram per square meter (g/m^2) | 112.40 (22.08) | 110.26 (23.92) | 115.59 (27.90) | 113.01 (24.18)
Left Ventricular Relative Wall Thickness [Mean (Standard Deviation); unit: proportion in hundredths] — Left ventricular relative wall thickness is measured as the ratio of the sum of the linear dimensions of the posterior wall and interventricular wall thicknesses in millimetres divided by the end-diastolic diameter of the left ventricular cavity in millimetres
  proportion in hundredths | 0.48 (0.07) | 0.49 (0.06) | 0.48 (0.08) | 0.48 (0.07)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: portion of volume in percent (%)] — The portion of blood volume ejected during the systole (stroke volume) in percent measured as the difference of end-diastolic and end-systolic volumes of left ventricle divided by end-diastolic volume of left ventricle using equations for biplane area-length method for two-dimensional echocardiographic measurements of left ventricular volume from 4- and 2-chamber imaging.
  portion of volume in percent (%) | 54.39 (6.32) | 54.77 (5.58) | 52.13 (6.12) | 53.79 (6.23)
Tricuspid Annular Plane Systolic Excursion [Mean (Standard Deviation); unit: millimeters] — Tricuspid annular plane systolic excursion assessed by M-mode echocardiography imaging in 4- and 2-chamber view by measuring the linear dimension of the displacement of the tricuspid annulus in millimetres relative to the right ventricular apex
  millimeters | 21.03 (2.77) | 20.88 (3.12) | 20.83 (2.21) | 20.95 (2.67)
Pulmonary Artery Systolic Pressure [Mean (Standard Deviation); unit: millimetres of mercury (mmHg)] — Pulmonary artery systolic pressure in millimetres of mercury (mmHg), estimated by Doppler-, echocardiography in the absence of right ventricular outflow tract obstruction or pulmonary stenosis, based on tricuspid regurgitant jet velocity using the modified Bernoulli equation and right atrial pressure measured by inferior vena cava diameter and collapsibility
  millimetres of mercury (mmHg) | 38.22 (8.67) | 36.67 (7.14) | 36.47 (7.77) | 37.47 (8.21)
Doppler- echocardiographic characteristics [Count of Participants; unit: Participants] — Number and percentage of study participants with specific qualitative doppler-echocardiographic characteristics of heart structure and function
  Participants
    Left ventricular hypertrophy | 115 | 34 | 68 | 217
    Increased left ventricular filling pressure | 23 | 6 | 18 | 47
    Right Ventricular Dilatation | 20 | 5 | 20 | 45
    Mitral annular calcification (MAC) | 9 | 3 | 9 | 21
    Secondary (functional) mitral regurgitation | 123 | 36 | 69 | 228
    Aortic valve calcification | 27 | 8 | 23 | 58
    Secondary (functional) aortic regurgitation | 24 | 17 | 41 | 82
    Secondary (functional) tricuspid regurgitation | 67 | 21 | 18 | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants Who Died From Any Cause (Death From Any Cause)
Description: The event of death from any cause reported by the physician according to the WHO Clinical criteria for the determination of death or the incident declared by the caregiver of the patient and checked for appropriateness in hospital registries or the national death registry within the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: Study participants of both sexes aged 35-79 years old, diagnosed with chronic coronary artery disease, who had undergone elective PCI and required P2Y12 inhibitor antiplatelet treatment
Measure: Count of Participants; unit: Participants
Groups:
- Normal Metabolizers of Clopidogrel: Study participants diagnosed with chronic coronary artery disease who had undergone elective PCI, tested with CYP2C19 genotyping and identified as NFA *2, *3 carriers. CYP2C19 Genotype-Guided Clopidogrel Treatment Clopidogrel as a component of preventive antiplatelet treatment, such as double antiplatelet treatment (DAPT), or an antiplatelet drug (clopidogrel) combined with the non-vitamin K antagonist oral anticoagulants (NOAC), incl. triple antiplatelet treatment (Aspirin, Clopidogrel and a NOAC), or antiplatelet monotherapy (Clopidogrel)
- Passive Metabolizers of Clopidogrel: Study participants diagnosed with chronic coronary artery disease who had undergone elective PCI, tested with CYP2C19 genotyping were identified as LoF *2, *3 allele carriers. CYP2C19 Genotype Guided Antiplatelet Treatment alternative to clopidogrel in conventional dosing regimen, as a component of preventive antiplatelet treatment, such as double antiplatelet treatment (DAPT) with ticagrelor or prasugrel, or prasugrel combined with the nonvitamin K antagonist oral anticoagulants (NOAC), or antiplatelet monotherapy (ticagrelor or prasugrel).
- Unspecified Metabolizers of Clopidogrel: Study participants diagnosed with chronic coronary artery disease who had undergone elective PCI were allocated to the arm through the randomisation, without CYP2C19 genotyping and clopidogrel metabolism phenotype was not specified
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 8 | 2 | 7

2. Primary Outcome: Number of Study Participants Who Died From Any Cardiovascular Cause (Death From Cardiovascular Cause)
Description: The event of death from any cardiovascular cause reported by the physician according the SCTI (Standardized Data Collection for Cardiovascular Trials Initiative) definitions or the incident declared by the caregiver of the patient and checked for appropriateness in hospital registries or the national death registry within the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 5 | 1 | 6

3. Primary Outcome: Number of Study Participants Who Died From Non-cardiovascular Causes (Death From Non-cardiovascular Cause)
Description: The event of death from a non-cardiovascular cause reported by the physician or the incident declared by the caregiver of the patient and checked for appropriateness in hospital registries or the national death registry within the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 3 | 1 | 1

4. Secondary Outcome: Number of Study Participants Who Experienced Non-fatal Myocardial Infarction (Non-fatal Myocardial Infarction)
Description: The clinical event of the non-fatal myocardial infarction detected during the study follow-up period and assessed by the 2012 Third Universal Definition of Myocardial Infarction as recommended by the SCTI (Standardized Data Collection for Cardiovascular Trials Initiative) definitions during the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Unspecified Metabolizers of Clopidogrel: Study participants diagnosed with chronic coronary artery disease who had undergone elective PCI were allocated to the arm through the randomisation, without CYP2C19 genotyping, and clopidogrel metabolism phenotype was not specified
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 4 | 1 | 4

5. Secondary Outcome: Number of Study Participants Who Experienced Unstable Angina or Angina Requiring Hospitalization (Unstable Angina)
Description: The clinical event corresponding to the unstable angina, or angina that requires hospitalization detected during the study follow-up period and assessed by the SCTI (Standardized Data Collection for Cardiovascular Trials Initiative) definitions during the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 14 | 3 | 16

6. Secondary Outcome: Number of Study Participants Who Experienced a Stroke or Transitory Cerebral Ischemic Event Within the Study Follow-up Period (Stroke or TIA)
Description: The clinical event of the stroke or transitory ischemic attack detected during the study follow-up period and assessed by the SCTI (Standardized Data Collection for Cardiovascular Trials Initiative) definitions for Stroke and Transient Ischemic Attack during the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 5 | 1 | 3

7. Secondary Outcome: Number of Study Participants Who Experienced Major Bleeding (Major Bleeding)
Description: The clinical event of major bleeding detected during the study follow-up period and assessed by the ARC-HBR (Academic Research Consortium for High Bleeding Risk) definitions as BARC type 3, 5 of bleeding during the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 3 | 2 | 4

8. Secondary Outcome: Number of Study Participants Who Experienced Non-major Bleeding (Non-major Bleeding)
Description: The clinical event of major bleeding detected during the study follow-up period and assessed by the ARC-HBR (Academic Research Consortium for High Bleeding Risk) definitions as BARC type 1 of bleeding during the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 2 | 4 | 4

9. Secondary Outcome: Number of Study Participants Who Experienced Heart Failure Event (Heart Failure Event)
Description: The clinical event of heart failure that requires hospitalization detected during the study follow-up period and assessed by the SCTI (Standardized Data Collection for Cardiovascular Trials Initiative) definitions during the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 14 | 4 | 9

10. Secondary Outcome: Number of Study Participants Who Experienced Percutaneous Coronary Intervention or Coronary Artery Bypass-grafting (Repeated Coronary Revascularization)
Description: The clinical event of any repeated coronary revascularization: percutaneous coronary intervention or coronary artery bypass-grafting detected during the study follow-up period and assessed by the SCTI (Standardized Data Collection for Cardiovascular Trials Initiative) definitions during the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 17 | 4 | 16

11. Other Pre Specified Outcome: Number of Study Cases in Each Arm With a Composite of Death From Any Cause, Non-fatal Myocardial Infarction, Stroke/TIA, or Major Bleeding Within the Study Follow-up (Net Adverse Clinical Events - NACEs)
Description: Net adverse clinical event (NACE) is assessed via measuring and putting together death from any cause, non-fatal myocardial infarction, stroke/TIA, or major bleeding (BARC type 3, 5) as potential outcomes for every studied case during the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 20 | 6 | 18

12. Other Pre Specified Outcome: Number of Study Cases in Each Study Arm With a Composite of Death From Any Cause, Myocardial Infarction, or Stroke/TIA Within the Study Follow-up (Major Adverse Cardiac or Cerebral Events - MACCEs)
Description: Major adverse cardiac or cerebral event (MACCE) is assessed by measuring and putting together death from cardiovascular cause, non-fatal myocardial infarction, or stroke/TIA as potential outcomes for every studied case during the study follow-up period, from the date of study enrollment until the date of the event.
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 142 | 38 | 70
Participants | 17 | 4 | 14

13. Other Pre Specified Outcome: Number of Study Cases With Certain Antiplatelet Treatment Selection (Dual Antiplatelet Treatment, Triple Antiplatelet Treatment, Combined Antiplatelet and Anticoagulant, or Antiplatelet Monotherapy) in Each Study Arm
Description: The number and percentage (%) of each arm of study participants treated with dual antiplatelet treatment, triple antiplatelet treatment, antiplatelet and non-vitamin K antagonist oral anticoagulant combination, or antiplatelet monotherapy
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 157 | 43 | 83
Participants
  Dual Antiplatelet Treatment (DAPT) | 114 | 27 | 72
  Triple antiplatelet treatment | 22 | 0 | 11
  Combined antiplatelet and non-vitamin K antagonist oral anticoagulant (NOAC) | 14 | 10 | 0
  Antiplatelet monotherapy | 7 | 6 | 0

14. Other Pre Specified Outcome: The Number of Study Cases With Certain Antiplatelet Medication (Aspirin, Clopidogrel, P2Y12 Inhibitor, Alternative to Clopidogrel, or A Non-vitamin K Antagonist Oral Anticoagulant (NOAC)) Prescription
Description: The number and percentage (%) of study participants treated with a certain antiplatelet drug - aspirin, clopidogrel, P2Y12 inhibitor alternative to clopidogrel, or a non-vitamin K antagonist oral anticoagulant (NOAC) in each study arm
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 157 | 43 | 83
Participants
  Aspirin | 136 | 32 | 83
  Clopidogrel | 157 | 0 | 83
  P2Y12 inhibitor, alternative to Clopidogrel | 0 | 38 | 0
  Non-vitamin K antagonist oral anticoagulant (NOAC) | 36 | 10 | 11

15. Other Pre Specified Outcome: The Number of Study Cases With Lipid-lowering Medication (Statin, or Combination With Ezetimibe, or Ezetimibe and PCSK9i) Prescription
Description: The number and percentage (%) of study participants treated with lipid-lowering medication - statin, or combined statin and ezetimibe, or statin, ezetimibe and PCSK9i in each study arm
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 157 | 43 | 83
Participants
  Statin | 87 | 27 | 21
  Combined statin and ezetimibe | 67 | 16 | 62
  Combined statin, ezetimibe and PCSK9i | 3 | 0 | 0

16. Other Pre Specified Outcome: The Number of Study Cases With Hypoglycemic Medication Prescription
Description: The number and percentage (%) of study participants treated with certain hypoglycemic medication - insulin, sodium-glucose cotransporter-2 (SGLT2) inhibitor, metformin, glucagon-like peptide-1 (GLP-1) receptor agonist, or dipeptidyl peptidase IV (DPP IV) inhibitor in each study arm
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 157 | 43 | 83
Participants
  Insulin | 4 | 2 | 4
  Sodium-glucose cotransporter-2 (SGLT2) inhibitor | 81 | 23 | 43
  Metformin | 39 | 12 | 31
  Glucagon-like peptide-1 (GLP-1) receptor agonist | 3 | 0 | 0
  Dipeptidyl peptidase IV (DPP IV) inhibitor | 31 | 10 | 30

17. Other Pre Specified Outcome: The Number of Study Cases With Other Common Evidence-Based Medication Prescription for Cardiovascular Risk Reduction
Description: The number and percentage (%) of study participants treated with other common evidence-based medication for cardiovascular risk reduction - angiotensin converting enzyme inhibitor (ACEi), angiotensin receptor blocker (ARB), angiotensin receptor neprilysin inhibitor (ARNi), beta adrenergic blocker, loop diuretic, mineralocorticoid receptor antagonist (MCRA), thiazide diuretic, calcium channel blocker, anti-arrhythmic drug or ivabradine in each study arm
Time Frame: within a 12-month of the study follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
Number analyzed (Participants) | 157 | 43 | 83
Participants
  Angiotensin converting enzyme inhibitor (ACEi) | 47 | 13 | 51
  Angiotensin receptor blocker (ARB) | 83 | 22 | 24
  Angiotensin receptor neprilysin Inhibitor (ARNi) | 21 | 7 | 20
  Beta adrenergic blocker | 129 | 34 | 80
  Loop diuretic | 43 | 8 | 31
  Mineralocorticoid receptor antagonist (MCRA) | 47 | 15 | 26
  Thiazide diuretic | 32 | 5 | 37
  Calcium channel blocker | 58 | 13 | 32
  Anti-arrhythmic drug | 22 | 11 | 3
  Ivabradine | 4 | 1 | 0

18. Other Pre Specified Outcome: Number of Study Participants Who Reported Their Health Status as Good or Satisfactory; or With the Appearance of CVD Symptoms; or With a Significant Inability to Self-care (Patient-Reported Health Status)
Description: The health status reported by the patient as: a) good or satisfactory; b) with the appearance of CVD symptoms; c) a significant inability to self-care ranked with severity degree of patient well-being, symptom burden, or ability for self-care, which is assessed according to the routine health related quality of life questionnaire definitions.
Time Frame: at 3, 6 and 12-month of the study follow-up
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Number of Study Participants Self-reported Angina Not Required Hospitalization (Patient-Reported Angina Not Required Hospitalization)
Description: The participant-reported last week episode of chest pain, or any discomfort, shortness of breath, or tightness in the chest due to angina not required hospitalization assessed by the CROQ (Coronary Revascularization Outcome Questionnaire) definitions.
Time Frame: at 3, 6 and 12-month of the study follow-up
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Number of Study Participants Reported Last Week's Shortness of Breath Due to Heart Failure Not Requiring Hospitalization (Patient-Reported Heart Failure Severity)
Description: The participant reported last week's shortness of breath due to mild physical activity or at rest not requiring hospitalization assessed by the PROMIS®-Plus-HF (Patient-Reported Outcomes Measurement Information System®-Plus-Heart Failure) profile definitions.
Time Frame: at 3, 6 and 12 months of the study follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12-month period of the study follow-up
Description: The data for adverse events were collected from the 250 participants who completed the study.
  The study routinely collects information on Major Adverse Cardiovascular and Cerebrovascular Events (MACCEs) that are severe in terms of their outcome and considered as clinical endpoints of the study. They are presented in the study outcomes section as well.
Groups:
- Unspecified Metabolizers of Clopidogrel: Study participants diagnosed with chronic coronary artery disease who had undergone elective PCI were allocated to the arm through the randomisation, without CYP2C19 genotyping and clopidogrel metabolism phenotype has not been specified
Arm/Group | Normal Metabolizers of Clopidogrel | Passive Metabolizers of Clopidogrel | Unspecified Metabolizers of Clopidogrel
All-Cause Mortality (participants affected / at risk) | 8/142 | 2/38 | 7/70
Serious Adverse Events (participants affected / at risk) | 23/142 | 10/38 | 25/70
Other Adverse Events (participants affected / at risk) | 4/142 | 4/38 | 5/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Metabolizers of Clopidogrel (N=142) | Passive Metabolizers of Clopidogrel (N=38) | Unspecified Metabolizers of Clopidogrel (N=70)
Major Bleeding (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 4 (4) — A bleeding event, mostly GI, classified as Type 2 or 3 by the BARC (Bleeding Academic Research Consortium) scale
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2) — Decrease in platelet count <100×109/L or <50% compared to the previous measurement assessed by complete blood count
Non-fatal Myocardial Infarction (Cardiac disorders) | 4 (4) | 1 (1) | 4 (4) — The clinical event of the non-fatal myocardial infarction detected during the study follow-up period and assessed by the 2012 Third Universal Definition of Myocardial Infarction
Unstable Angina or Angina Requiring Hospitalization (Cardiac disorders) | 8 (14) | 3 (3) | 10 (16) — The clinical event corresponding to the unstable angina, or angina that required hospitalization, detected during the study follow-up period and assessed by the Standardized Data Collection for Cardiovascular Trials Initiative (SCTI) definitions
Stroke or Transitory Cerebral Ischemic Event (Vascular disorders) | 5 (5) | 1 (1) | 3 (3) — The clinical event of the stroke or transitory ischemic attack detected during the study follow-up period and assessed by theStandardized Data Collection for Cardiovascular Trials Initiative (SCTI) definitions
Heart Failure Event (Cardiac disorders) | 1 (14) | 2 (4) | 2 (9) — The clinical event of heart failure that requires hospitalization detected during the study follow-up period and assessed by the Standardized Data Collection for Cardiovascular Trials Initiative (SCTI) definitions
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Metabolizers of Clopidogrel (N=142) | Passive Metabolizers of Clopidogrel (N=38) | Unspecified Metabolizers of Clopidogrel (N=70)
Minor bleeding (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 4 (4) — Any bleeding event classified as Type 1 by BARC (Bleeding Academic Research Consortium) scale, bleeding from gums, nosebleeds, or prolonged bleeding from cuts, did not seek unplanned medical attention
Skin Rashes and Itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) — Skin Rashes and Itching as the manifestation of hypersensitivity or allergy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT06665919/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT06665919/ICF_001.pdf